CLINICAL TRIAL: NCT05826691
Title: Impact of Prostate Surgery for LUTS on Patients' QOL With Emphasis on Sexual- and Ejaculatory Function
Brief Title: Benign Prostate Surgery and QOL and Sexual Function
Acronym: BEPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: TC Erciyes University (Other); Gaziosmanpasa Research and Education Hospital (Other Government); Goztepe Training and Research Hospital (Other); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Ankara Education and Research Hospital (Other Government); Uludag University (Other); Kırıkkale University (Other); SB Istanbul Education and Research Hospital (Other); Kayseri City Hospital (Other Government); Bagcilar Training and Research Hospital (Other Government); Ataturk University (Other); Sisli Hamidiye Etfal Training and Research Hospital (Other); Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other); Haydarpasa Numune Training and Research Hospital (Other); SBÜ Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi (Other); Fatih Sultan Mehmet Training and Research Hospital (Other); Firat University (Other); Recep Tayyip Erdogan University (Other); Yuzuncu Yil University (Other); Ondokuz Mayıs University (Other); Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government); Ankara City Hospital Bilkent (Other); Izmir Katip Celebi University (Other); Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, vahit guzelburc, Assistant Professor of Urology, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-2928
Record Dates: First submitted 2023-03-22; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Quality of Life; Sexual Dysfunction; Ejaculatory Dysfunction; Lower Urinary Tract Symptoms; Erectile Dysfunction; Incontinence
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Ejaculatory Dysfunction; Lower Urinary Tract Symptoms; Erectile Dysfunction | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients required prostate surgery for LUTS: Patients with LUTS attributable to bladder outlet obstruction because BPH
  Interventions: Procedure: Monopolar / Bipolar Transurethral resection of prostate (TURP), photovaporisation (PVP), Plasmakinetic (PK), Holmium laser enucleation of the prostate (HOLEP) or open prostatectomy (OP)).

INTERVENTIONS:
Procedure: Monopolar / Bipolar Transurethral resection of prostate (TURP), photovaporisation (PVP), Plasmakinetic (PK), Holmium laser enucleation of the prostate (HOLEP) or open prostatectomy (OP)). — Any procedure advised by the EAU guidelines to ovrecome bladder outlet obstruction
  Other Names: Open prostatectomy

SUMMARY:
Rationale: A variety of surgical techniques have been described for surgical treatment of male LUTS because of BPH, which has different outcomes and may result in adverse events regarding ejaculatory function and erection, resulting in a negative impact on QOL on short- and mid-term follow-ups.

Objective: To compare outcomes of BPH surgery using a conventional versus ejaculation preserving technique on QOL-related aspects with emphasis on ejaculatory and erectile function.

Study design: This study is a prospective longitudinal multi-center trial to compare the ejaculatory and erectile function outcomes between conventional and ejaculation preserving BPH surgical procedures/techniques. Baseline characteristics will be recorded, as well as short and mid-term follow-up.

Study population: The study population comprises patients who will undergo BPH surgery in the participating centers.

Intervention: All patients will undergo BPH surgery (including but not restricted to Monopolar / Bipolar Transurethral resection of the prostate (TURP), photo vaporisation (PVP), Plasmakinetic (PK), Holmium laser enucleation of the prostate (HOLEP) or open prostatectomy (OP)).

Main study parameters/endpoints: Primary endpoint is to compare the baseline to the short-term (3 months) and mid-term (6 months) ejaculation function and QoL outcomes. The secondary endpoint is the short and mid-term erection function and QoL outcomes compared to baseline.

Nature and extent of the burden and risks associated with participation, benefit, and group relatedness: Patients' burden and risk associated with participating in this trial do not differ among surgical procedures or techniques used. In all groups, patients will undergo a BPH surgery and will be followed for six months at 3 visits.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a common condition in aging men, which may lead to lower urinary tract symptoms (LUTS) and sexual dysfunction, negatively impacting the patients' quality of life. Despite allowing relief from LUTS, classical medical and surgical treatments for BPH have always been burdened by important consequences on the patients' sexual and ejaculatory function. Over the past three decades, research has focused on the development of new surgical strategies to reduce morbidity and complications of surgical procedures, however, in most cases overlooking the impact on the patients' quality of life aspects.

Despite the well-documented advantages of Laser techniques over transurethral resection of prostate (TURP) and open prostatectomy (OP), they have not been able to overcome postoperative ejaculatory dysfunction (EjD). It is well known that loss of ejaculation after endoscopic surgery was and is still attributed by many to compromising the ejaculatory mechanism, causing retrograde ejaculation. The ejaculatory mechanism has long been misunderstood and misinterpreted. However, recent evidence on ejaculation physiology has demonstrated the importance of the tissues surrounding the verumontanum, rather than the bladder neck, for outward ejaculation . Dynamic transrectal ultrasonography (TRUS) has shown how, just before ejaculation, the verumontanum undergoes a caudal shift, contacting the anterior wall of the urethra, allowing the antegrade progression of semen, which is emitted into the inframontanal urethra and expelled, almost simultaneously, through the external sphincter. No accumulation of semen inside the prostatic urethra, and therefore, generation of a high-pressure area was demonstrated. A fundamental role in this process is played by the musculus ejaculatorious, a longitudinal strain of muscle fibers, which originate from around the ejaculatory ducts and extend caudally in the urethral crest, inserting below the urethral sphincter. Contraction of the musculus ejaculatorious could be responsible not only for the emission of semen from the ejaculatory ducts into the prostatic urethra, but also for the correct movement of the veru montanum during ejaculation. Based on these findings, supramontanal and paracollicular tissue-sparing surgical techniques have been developed. Ejaculation preserving (EP) techniques have been applied to TURP, Photoselective vaporization of the prostate (PVP) and Holmium laser enucleation of the prostate (HOLEP) with encouraging results.

EP technique will be performed as:

During BPH open and endoscopic surgery, all prostatic tissue except adjacent to the verumontanum is removed. Ejaculation preserving endoscopic prostatectomy is a new technique, where all apical prostatic tissue is removed by resecting tissue up to 1 cm above the verumontanum laterally and proximally, to preserve antegrade ejaculation.

Operating physicians will report the type or surgery technique in terms of preservation or not of the ejaculation as: "no", "probably no", "probably yes" or "yes"

This study aims to compare the impact of different BPH surgical techniques on QOL by using subjective and objective tools to better demonstrate short- and mid-term outcomes.

Quality of Life related outcomes, (ejaculatory and erectile functions will be assessed by Patients Related outcomes (PROs). The following culturally validated questionnaires will be distributed to the patients at baseline and in the follow-up controls after surgery.

- ShortForm-12 (SF-12)

Consist of 12 generic qualty of life (QOL) questions, scores range between 12-56. The higher scores are associated with QOL.

- International Index of Erectile Function-5 (IIEF-5):

Consist of 5 questions. Each question scores 1-5, in total scores range between 5-25. The lower scores are associated with with worse erectile function

- Male Sexual Health Questionnaire-Ejaculatory Dysfunction-Short Form (MSHQ-EjD-SF)

Consist of 3 questions for ejaculatory function and 1 question for difficuty in ejaculation. Each question scores 0-5. The higher scores are associated with worse function.

- International Prostate Symptoms Score (IPSS)

Consist of 7 lower urinary tract symptoms (LUTS) and 1 quality of life questions (QOL). Each LUTS question scores 0-5, in total scores range between 0-35. The higher scores are associated with worse symptoms. QOL question scores 0-6 and the higher score are associated with lower qualty of life.

-Modified Clavien-Dindo grading system for asessment of adverse events and compliacations.

Consist of 5 questions (Question 3 and 4 have 2 subgroubs as a and b). Grade 1 is the minor complication without the need for phamacological treatment or surgical, endoscopic and radiologic interventions. Grade 5 (The highest score) is defined as 'Death of a patient'

Study design This study is a prospective longitudinal multi-center study in which the ejaculation and erection function as well as QoL aspects after BPH surgery for male LUTS are compared between traditional versus ejaculation preserving approach. Each participating center chooses and performs a BPH surgical procedure (TURP, PVP, HOLEP, OP) with or without an ejaculation preserving technique to their discretion. Data from all participating centers will be collected through electronic Case Report Forms (eCRFs), with use of an online Data Management System (DMS), which is located and maintained at Istanbul Medipol University. Faculty in the Division of Biostatistics and Health Informatics at Istanbul Medipol University will perform all data quality checks, analyses and reporting.

Population The study population comprises males (aged >40 years) presenting with lower urinary tract symptoms (LUTS) and eligible for BPH operation. All participating institutions are expert centers where secondary/tertiary health care is provided.

Perioperative complications will be graded according the Dindo-Clavien classification

The investigators will assess the objective success of the different interventions by means of Uroflowmetry.

Follow up schedule: patients will be controlled post-operatively by 2 follow-up visits (6-12 week and 6 months)

Data collection and quality control:

Pertinent patient data from all participating centers will be centrally collected through electronic Case Report Forms (eCRFs) through an online Data Management System (DMS), located and maintained at Istanbul Medipol University. Patients will be pseudonymized and only the corresponding PIs in the different Institutions will have access to the identity if necessary.

The Division of Biostatistics and Health Informatics at Istanbul Medipol University will monitor data collection and perform data quality checks, analysis and reporting.

Sample calculation:

The investigators hypothesized that conventional BPH surgical procedures will result in around 1-unit decrease in ejaculation function at 6-month evaluation with respect to baseline (mean normalized scores for age and country) while the ejaculation preserving BPH surgical

procedures will retain the ejaculation function unchanged. In QoL at least 3 units differential improvement are expected with respect to the mean baseline scores at 6-months between the ejaculation preserving and the conventional techniques.

When considering both co-primary objectives a total sample of 1120 participants will be sufficient to detect the differences. By considering an attrition rate of 25% at 6-month, the total enrollment is planned at 1500 participants, of whom around 300 are anticipated to undergo ejaculation preserving BPH surgeries according to previous experience and literature.

Statistical analysis

Primary objective measures will be analysed using an Analysis of Covariance (ANCOVA) framework where baseline measures and peri- and post-surgery characteristics will be added to the model as covariates, the changse in the co-primary objectives measure from baseline to 6-months as the dependent variable, and the study arm being the primary predictor. In these models, interaction between Study Arm and patient and BPH surgery characteristics will also be investigated. To satisfy the model assumptions, data-transformation approaches such as log-transformation may be applied to the outcome measures as well as the predictors as necessary.

As part of the secondary objectives, surgery-specific subset analysis will be conducted using the ANCOVA approach if available data allows and supports such subset analysis.

Complications and Adverse Events will be described as proportions and compared between the two-arms of the study using Chi-Square or Fisher's exact test and Logistic Regression with baseline measures and peri- and post-surgery characteristics added to the model as covariates as scientifically justified. Poisson regression will be used for repeat events and complications.

The study is designed and will follow the ethical principles for medical research involving human subjects of the Helsinki Declaration of October 2013 (https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/)

Summary of known and potential risks and benefits Follow-up and controls will not differ from the patients control arm in the study.The risks that patients are subject to in this trial do not differ from risks associated with conventional surgery without specific intention to preserve ejaculation. Patients will receive the standard treatment in addition to the extra care that is provided to them in the framework of this study.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent
* Is aged 40 years or older
* With or without erectile function and/or antegrade ejaculation
* No limitation for prostate volume
* Height 150-250 cm
* Weight 40-150 kg
* Age 40-90 years old
* PSA 0.1-30 ng/ml
* Creatinine 0.5-4mg/dl

Exclusion Criteria:

* History of BPH surgery

  * History of pelvic radiation
  * History of chronic prostatitis or chronic pelvic pain syndrome
  * History of urethral stricture
  * History of bladder neck contracture
  * Has or has had tumors in the urinary tract
  * Has or has had prostate cancer
  * Has had previous irradiation of the pelvis
  * Has bladder stone
  * Has urinary tract infection (UTI)
  * Has chronic UTI
  * Has neurogenic disorder
  * Has conditions associated with a risk of poor protocol compliance
  * Has participation in other clinical studies with investigational drugs either concurrently or within the last 30 days

Ages: 40 Years to 90 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Because of the nature of prostatic obstruction only males or individuals with prostate gland can be included
Study Population: Adult male patients, complaining of LUTS who require surgery because BPH
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Preservation of QOL after surgery for BPH | Baseline to 6 months after surgery
  QOL will be assessed before and after by means of validated SF-12 questionnaire
Preservation of sexual function after surgery for BPH | Baseline to 6 months after surgery
  Sexual function will be assessed before and after by means of IIEF-5 validated questionnaire
Preservation of ejaculatory function after surgery for BPH | Baseline to 6 months after surgery
  Ejaculatory function will be assessed before and after by means of MSHQ-EjD-SF validated questionnaire
Preservation of voiding function after ejaculation preserving BPH surgery | Baseline to 6 months after surgery
  LUTS will be assessed before and after by means of IPSS validated questionnaire

SECONDARY OUTCOMES:
Comparison of post-operative complications among the different disobstructive methods | From the day of the operastion up to 90 days
  Adverse events/complications will be recorded by using Modified Dindo-Clavien for urological surgery
Comparison objective outcomes of uroflowmetry Qmax parameter (ml/sec) in relation to outcomes in preservation of ejaculation and unpreserved surgery | Baseline to 6 months after surgery
  Pre- and postoperative uroflowmetry maximum flow rate (Qmax; ml/sec) parameter will be compared between ejaculation preserved and ejaculation not preserved operations
Comparison residual urine volumes (Post-voided residual urine, ml) by ultrasound measurement in relation to outcomes in preservation of ejaculation and unpreserved surgery | Baseline to 6 months after surgery
  Pre- and post-operative residual urine volume (PVR, ml) will be assessed by ultrasound will be compared between ejaculation preserved and ejaculation not preserved operations
Comparison changes in erectile function between conventional and preserving ejaculatory techniques by using IIEF-5 validated questionnarie | Baseline to 6 months after surgery
  Pre- and postoperative erectile function will be compared between conventional and preserving ejaculatory

CONTACTS AND LOCATIONS:
Overall Officials: Johan J de la Rosette, MD PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No